CLINICAL TRIAL: NCT03833934
Title: ALCMI-011: Study of Plasma Next Generation Sequencing for Assessment, Characterization, Evaluation of Patients With ALK Resistance (SPACEWALK)
Brief Title: Study of Plasma NGS for Assessment, Characterization, Evaluation of Patients With ALK Resistance
Acronym: SPACEWALK
Status: Completed | Type: Observational
Sponsor: Addario Lung Cancer Medical Institute (Other)
Collaborators: Dana-Farber Cancer Institute (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ALCMI-011; 5R21CA234816 (NIH)
Record Dates: First submitted 2019-01-28; First posted 2019-02-07 (Actual); Results first posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: ALK positive
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood specimens will be tested for genetic mutations in ALK and other genes that may be important for lung cancer. The participant and their doctor will receive a copy of the test results. The test results will describe the gene alterations that are detected in the blood sample. The assay covers a region of the ALK gene and other lung cancer genes where resistance alterations can occur.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ALK-positive NSCLC with progression: Patients in this group signed consent, met eligibility criteria, and all had ALK-positive cancer of a primary lung lesion with systemic progression (excluding the central nervous system)

SUMMARY:
ALK-positive lung cancer is a subtype of lung cancer which carries a change in a gene called ALK (anaplastic lymphoma kinase). There are now many drugs for patients with ALK-positive lung cancer that slow cancer growth. However, after some time, just as bacteria evolve resistance to antibiotics, ALK-positive lung cancers evolve ways to avoid the therapies by developing new mutations so the drugs lost their effectiveness. These new mutations can potentially be treated with a different drug. For these new therapies, the range of mutations that can develop at resistance is not well understood.

It is now possible to detect the presence of mutations or changes in the genetic structure in lung cancer by analyzing a patient's blood for bits of material shed by tumor. This approach is often called a liquid biopsy. Recently, researchers have shown that looking at tumor molecules through liquid biopsies can provide doctors with some of the same information that tissue biopsies provide. For example, liquid biopsies can be used to detect mutations that cause drug resistance. Obtaining liquid biopsies on patients with ALK-positive lung cancers at resistance to therapy may help better understand the different mutations that develop and guide therapy decisions.

In this research study, a blood specimen will be collected and submitted for liquid biopsy analysis at a commercial diagnostic company. This company specializes in analyzing tumor material found in blood. Specifically, it will look for genetic changes in the ALK gene that could help understand why a cancer has developed drug resistance.

This research study is for lung cancer patients with ALK-positive lung cancer who had been on a newer ALK targeted treatment (such as ceritinib, alectinib, brigatinib, or lorlatinib) to determine whether they have developed ALK resistance mutations. The investigators will collect a blood sample to examine these mutations. Participants will not have to have a tissue biopsy to participate in this study. Participants do not have to visit Dana-Farber Cancer Institute (DFCI) to participate. All study procedures will be performed remotely.

DETAILED DESCRIPTION:
SPACEWALK is an innovative remote consent and participation study using next-generation sequencing (NGS) of plasma cell-free DNA (cfDNA) to characterize resistance mechanisms arising in ALK-positive non-small cell lung cancer (NSCLC) after progression while on a next generation ALK tyrosine kinase inhibitor (TKI). Additionally, the study will capture the potential of genomic-driven resistance therapy approach for effecting outcomes in patients with advanced ALK-positive NSCLC and TKI resistance. Finally, the study will assess the role of repeat plasma NGS in evaluating drug response.

The study will accrue patients with advanced ALK-positive NSCLC on systemic progression (outside the brain) while on treatment with a next-generation ALK TKI. Any patient interested in the study will find information about the study on the study website. The patient will consent remotely through the study website and documentation of advanced ALK-positive NSCLC and systemic progression while on a next-generation ALK TKI. The study team will reach out to the patient to confirm eligibility and send a blood collection kit. In the study kit the study participants will find all the necessary materials for local blood draws, and collected specimens will be sent directly to the central study laboratory (Resolution Bioscience) for plasma NGS.

Plasma NGS of cfDNA will involve sequencing of 19 genes, including ALK, permitting remote tumor genotyping. Plasma NGS analysis and results will be done following standard procedures of the Resolution Bioscience CLIA-certified laboratory. Results will be sent to study participants, their physicians and study team within 1-2 weeks. Plasma NGS reports will not include any specific treatment recommendations but will describe the presence of an ALK rearrangement, ALK resistance mutation, or other relevant mutations.

Study participants are followed remotely. The study coordinator will contact the participants weekly for 4 weeks after enrolled into the study to learn of any new treatment initiation and to release an additional plasma collection kit 2-4 weeks after starting treatment. Study participants will then be remotely contacted every 3 months to follow clinical outcomes on therapy for up to 2 years. If the cancer progresses on the participant's new treatment, the patient will have the option to provide a third blood specimen. Medical records and local imaging will be collected and studied.

The primary objective of the study is to characterize ALK TKI resistance to next-generation ALK TKIs in patients with advanced ALK-positive NSCLC. Secondarily, the investigators will assess the potential of plasma NGS to impact outcome on treatment by studying time to treatment discontinuation. Serial plasma NGS will also be assessed as a response biomarker. A total of 300 patients are planned to be enrolled, with the expectation that approximately 200 will have tumor-related mutations detected in plasma NGS.

ELIGIBILITY:
Inclusion Criteria:

* Men or women older than 18 years at the time of consent.
* Demonstration of having advanced ALK positive NSCLC.
* Systemic progression (not CNS only progression) within the past 30 days while receiving a next generation ALK TKI.
* Patient must not have started a new line of therapy before signing the informed consent form.
* Willingness to provide a blood specimen prior to the initiation of a new line of treatment.
* Willing to provide clinical and medical information to the study team as required.
* Ability to read, write and communicate in English.
* Ability to sign a web-based informed consent form.

Exclusion Criteria:

* Participants who are unable to provide informed consent.
* Participants who are 18 years of age or younger.
* Participants who are unable to comply with the study procedures.
* Known existence of an uncontrolled intercurrent illness including, but not limited to, psychiatric illness or social situations that would impair compliance with study requirements.
* Participants who have previously enrolled to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This research study is for lung cancer patients with ALK-positive lung cancer who had been on a newer ALK targeted treatment (such as ceritinib, alectinib, brigatinib, or larlatinib).
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2019-01-23 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey R Oxnard, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lawrence MN, Tamen RM, Martinez P, Sable-Hunt A, Addario T, Barbour P, Shaffer T, Hosseini SA, Bertucci C, Lim LP, Hong F, Michael K, Simon GR, Riess JW, Awad MM, Oxnard GR. SPACEWALK: A Remote Participation Study of ALK Resistance Leveraging Plasma Cell-Free DNA Genotyping. JTO Clin Res Rep. 2021 Feb 3;2(4):100151. doi: 10.1016/j.jtocrr.2021.100151. eCollection 2021 Apr. PMID 34590008

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were referred by means of their treating physician or social media to a study website (https://alcmi.net/research/spacewalk-study/) and completed a contact form indicating their interest in participating in the study and answered a prescreening questionnaire. If the patients indicated they have ALK-positive NSCLC and are progressing on an ALK TKI, they were contacted by the study staff who then released access to an online consent form to the patient.
Period: Overall Study
Arm/Group | ALK-positive NSCLC With Progression
Started | 62
Completed | 62
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | ALK-positive NSCLC With Progression
Number analyzed (Participants) | 62
Age, Continuous [Median (Full Range); unit: years] | 55 [21 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 40
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants] — Region of Enrollment, Study conducted in United States
  participants
    United States | 62
Subjects diagnosed with Advanced ALK positive NSCLC with progression [Number; unit: participants] | 62

OUTCOME MEASURES:

1. Primary Outcome: Prevalence of ALK Fusion
Description: To determine the prevalence of the ALK gene fusion in the cohort of patients with ALK-positive NSCLC with progression
Time Frame: 32 months
Measure: Count of Participants; unit: Participants
Arm/Group | ALK-positive NSCLC With Progression
Number analyzed (Participants) | 62
Participants | 27

2. Primary Outcome: ALK Fusion Allelic Frequency
Description: To determine the relative percentage of the ALK fusion within the cohort's gene pool
Time Frame: 32 months
Population: Patients with detected ALK fusion
Measure: Median (Full Range); unit: percentage of the ALK fusion
Arm/Group | ALK-positive NSCLC With Progression
Number analyzed (Participants) | 27
percentage of the ALK fusion | 2.6 [0.1 to 37]

3. Primary Outcome: Overall Prevalence of ALK Resistance Mechanism Among Patients With the ALK Fusion
Description: To determine the overall prevalence of ALK resistance mechanism in patients with detectable ALK fusion in plasma as determined per plasma NGS
Time Frame: 32 months
Population: Patients with detected ALK fusion
Measure: Count of Participants; unit: Participants
Arm/Group | ALK-positive NSCLC With Progression
Number analyzed (Participants) | 27
Participants | 17

4. Primary Outcome: Type of Resistance Mechanism: One or More Secondary ALK Kinase Domain Resistance Mutations
Description: To determine the prevalence of the various types of ALK resistance mechanisms as measured by NGS
Time Frame: 32 months
Population: Patients with detected ALK fusion
Measure: Count of Participants; unit: Participants
Arm/Group | ALK-positive NSCLC With Progression
Number analyzed (Participants) | 27
Participants | 8

5. Primary Outcome: Type of ALK Resistance Mechanism: Both ALK Resistance Mutations and Bypass Resistance
Description: To determine the prevalence of the various types of ALK resistance mechanisms as measured by NGS
Time Frame: 32 months
Population: Patients with detected ALK fusion
Measure: Count of Participants; unit: Participants
Arm/Group | ALK-positive NSCLC With Progression
Number analyzed (Participants) | 27
Participants | 6

6. Primary Outcome: Prevalance of ALK Restance Mechanism: Bypass Track Resistance
Description: To determine the prevalence of the various types of ALK resistance mechanisms as measured by NGS
Time Frame: 32 months
Population: Patients with detected ALK fusion
Measure: Count of Participants; unit: Participants
Arm/Group | ALK-positive NSCLC With Progression
Number analyzed (Participants) | 27
Participants | 3

7. Secondary Outcome: Changed Treatment for NSCLC
Description: Initiated a new ALK tyrosine kinase inhibitor for treatment of NSCLC following enrollment in the study
Time Frame: 32 months
Population: Patients with at least 3 months of follow-up time
Measure: Count of Participants; unit: Participants
Arm/Group | ALK-positive NSCLC With Progression
Number analyzed (Participants) | 59
Participants | 49

8. Secondary Outcome: Treatment Outcome: >50% Reduction of ALK Fusion Allelle Frequency
Description: New ALK TKI treatment resulted in >50% reduction of ALK fusion allelle frequency
Time Frame: 32 months
Population: Patients who had additional optional blood draw following initiation of new ALK TKI therapy
Measure: Count of Participants; unit: Participants
Arm/Group | ALK-positive NSCLC With Progression
Number analyzed (Participants) | 14
Participants | 7

ADVERSE EVENTS:
Time Frame: Adverse event data not applicable for this study
Description: Adverse event data not applicable for this study
Arm/Group | ALK-positive NSCLC With Progression
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-15): https://cdn.clinicaltrials.gov/large-docs/34/NCT03833934/Prot_SAP_000.pdf